CLINICAL TRIAL: NCT02730234
Title: JetStream Atherectomy for the Treatment of In-stent Restenosis of the Femoropopliteal Artery
Brief Title: JetStream Atherectomy for the Treatment of In-stent Restenosis
Acronym: JET-ISR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Cardiovascular Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCRF-S-002-2015
Record Dates: First submitted 2016-03-25; First posted 2016-04-06 (Estimated); Results first posted 2021-01-29 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2020-10

CONDITIONS: Femoropopliteal In-stent Restenosis
MeSH Terms: interventions — Angioplasty, Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- JetStream XC with balloon angioplasty (Experimental): The intervention consists of JetStream atherectomy of femoropopliteal in-stent restenosis using the JetStream XC device followed by adjunctive balloon angioplasty in all patients.
  Interventions: Device: JetStream XC with balloon angioplasty

INTERVENTIONS:
Device: JetStream XC with balloon angioplasty — JetStream XC to treat femoropopliteal in-stent restenosis followed by adjunctive balloon angioplasty (same arm). The control arm in this study is historic.
  Other Names: JetStream Navitus

SUMMARY:
The purpose of this study is to test the hypothesis that Jetstream atherectomy (JS) and adjunctive balloon angioplasty (PTA) (JS +PTA) improves target lesion revascularization (TLR) at 6 months follow-up when compared to historic data from PTA alone in the treatment of femoropopliteal (FP) arterial In-stent restenotic (ISR) disease.

This is a prospective, multicenter, single arm study evaluating the investigational use of Jetstream Atherectomy (JS) and adjunctive balloon angioplasty (JS +PTA) in the treatment of FP ISR lesions in subjects with claudication or limb ischemia (Rutherford clinical category (RCC) of 2-4) (lesion length ≥ 4 cm). The comparator arm is historic data from plain old balloon angioplasty derived from a Meta-analysis of the 3 published randomized trials in the field.

DETAILED DESCRIPTION:
The Boston Scientific Jetstream XC catheter is a rotating, aspirating, expandable catheter for active removal of atherosclerotic disease and thrombus in peripheral vasculature. The JS XC System has been cleared by the Food and Drug Administration (FDA) for use in the peripheral vasculature to treat denovo and non-stent infrainguinal lesions

Several studies have shown that stenting of the FP artery leads to higher long term patency. Bare metal stents however have not shown conclusively to reducemTLR which is in contrast to drug coated balloons (DCB) and drug coated stents (DCS). Irrespective, stenting has several disadvantages including a continued high rate of restenosis and stent fractures that is progressive with time. FP ISR occurs in more than one third of patients at 1 year and up to 49% at 2 years. Complex lesions (long, Trans-Atlantic Inter-Society Consensus II C/D lesions, total occlusions), certain demographics (female gender, diabetes mellitus), critical limb ischemia and significant stent fractures are associated with a higher rate of restenosis. Also the majority of occluded stents are restenotic-thrombotic and generally are more challenging to treat.

Recently 3 randomized trials were presented in treating FP ISR; the EXCImer Laser Randomized Controlled Study for Treatment of FemoropopliTEal In-Stent Restenosis (EXCITE ISR) trial (randomized laser + PTA vs PTA alone), the RELINE trial (Propaten Bioactive Surface vs. standard balloon angioplasty for treatment of in-stent restenosis in the superficial femoral artery) and the Randomized Femoral Artery In-Stent Restenosis (FAIR) Trial. All these studies showed superiority over PTA in treating FP ISR. Early animal data (porcine model of FP ISR) and feasibility human data (JetStream ISR study) have shown that the JetStream device is effective in ablating restenotic tissue within restenotic FP stents and had no safety concerns within well apposed stents and in the absence of Class III and IV fractures.

The purpose of this study is to assess and estimate the effect of treating FP ISR with plaque excision using JS in combination with adjunctive PTA and compare this to historic control of PTA. The comparator arm is historic data from PTA derived from a study-level meta-analysis of the 3 published randomized trials in the field.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic peripheral arterial disease (Rutherford Becker Class II to IV)
2. Previously treated with stenting in the femoropopliteal segment
3. No limit on how many times the target in-stent restenotic lesion has been previously treated.
4. There is no exclusion based on how the prior treatment was done including if drug eluting balloons or stents have been used. Covered stents cannot be included
5. There is no limit on the length of the target lesion as long as only one target lesion is treated and enrolled

Exclusion Criteria:

Subjects must meet all of the following criteria to be eligible to participate in this study:

1. Subject is 18 years of age or older.
2. Subject presents with clinical evidence of peripheral arterial disease with ISR in the femoropopliteal segment (includes common femoral, superficial femoral and popliteal)
3. Subject presents with a Rutherford Classification of 2-4 and has symptoms of rest limb pain or claudication.
4. Target lesion(s) must be viewed angiographically and have ≥50% stenosis.
5. The atherectomy wire must be placed entirely across all lesions to be treated with no visible evidence of clear or suspected subintimal/substent wire passage.
6. The main target vessel reference diameter must be > or = 5 mm and ≤ 7 mm
7. One patent distal run-off vessel with <70% disease and with brisk flow is required.
8. Intraluminal crossing of the lesion. If this is not certain, IVUS may be used to verify this per operator's discretion
9. Patient has signed approved informed consent.
10. Patient is willing to comply with the follow-up evaluations at specified times.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04; Primary Completion 2020-02-04 (Actual); Study Completion 2020-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas W Shammass, MD, MS, Principal Investigator — Midwest Cardiovascular Research Foundation; Subhash Banerjee, MD, Principal Investigator — VAMC, Dallas, Texas
Locations (13):
- United States (13):
  - Eastern Colorado Healthcare System, Denver, Colorado
  - Florida Hospital Heartland Medical Center, Sebring, Florida
  - Advocate Health, Downers Grove, Illinois
  - Midwest Cardiovascular Research Foundation/Trinity Medical Center, Bettendorf, Iowa
  - Midwest Cardiovascular Research Foundation/Genesis Medical Center, Davenport, Iowa
  - Endovascular Technologies, LLC, Shreveport, Louisiana
  - Atlantic Medical Imaging, Galloway, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Promedica Toledo Hospital, Toledo, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - US Departmetn of Veterans Affairs, Oklahoma VA Medical Center, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - VA North Texas Health Care System: Dallas VA Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
Data will be shared in aggregate in a manuscript. No plan to share individual patient data

REFERENCES:
- [Background] Shammas NW, Aasen N, Bailey L, Budrewicz J, Farago T, Jarvis G. Two Blades-Up Runs Using the JetStream Navitus Atherectomy Device Achieve Optimal Tissue Debulking of Nonocclusive In-Stent Restenosis: Observations From a Porcine Stent/Balloon Injury Model. J Endovasc Ther. 2015 Aug;22(4):518-24. doi: 10.1177/1526602815592135. Epub 2015 Jun 24. PMID 26109627
- [Background] Krankenberg H, Tubler T, Ingwersen M, Schluter M, Scheinert D, Blessing E, Sixt S, Kieback A, Beschorner U, Zeller T. Drug-Coated Balloon Versus Standard Balloon for Superficial Femoral Artery In-Stent Restenosis: The Randomized Femoral Artery In-Stent Restenosis (FAIR) Trial. Circulation. 2015 Dec 8;132(23):2230-6. doi: 10.1161/CIRCULATIONAHA.115.017364. Epub 2015 Oct 7. PMID 26446728
- [Background] Beschorner U, Krankenberg H, Scheinert D, Sievert H, Tubler T, Sixt S, Noory E, Rastan A, Macharzina R, Zeller T. Rotational and aspiration atherectomy for infrainguinal in-stent restenosis. Vasa. 2013 Mar;42(2):127-33. doi: 10.1024/0301-1526/a000256. PMID 23485840
- [Background] Shammas NW, Shammas GA, Aasen N, Jarvis G. Number of Blades-up Runs Using JetStream XC Atherectomy for Optimal Tissue Debulking in Patients with Femoropopliteal Artery In-Stent Restenosis. J Vasc Interv Radiol. 2015 Dec;26(12):1847-51. doi: 10.1016/j.jvir.2015.08.026. PMID 26596178
- [Background] Shammas NW, Shammas GA, Banerjee S, Popma JJ, Mohammad A, Jerin M. JetStream Rotational and Aspiration Atherectomy in Treating In-Stent Restenosis of the Femoropopliteal Arteries: Results of the JETSTREAM-ISR Feasibility Study. J Endovasc Ther. 2016 Apr;23(2):339-46. doi: 10.1177/1526602816634028. Epub 2016 Feb 26. PMID 26921281
- [Background] Bosiers M, Deloose K, Callaert J, Verbist J, Hendriks J, Lauwers P, Schroe H, Lansink W, Scheinert D, Schmidt A, Zeller T, Beschorner U, Noory E, Torsello G, Austermann M, Peeters P. Superiority of stent-grafts for in-stent restenosis in the superficial femoral artery: twelve-month results from a multicenter randomized trial. J Endovasc Ther. 2015 Feb;22(1):1-10. doi: 10.1177/1526602814564385. PMID 25775672
- [Background] Dippel EJ, Makam P, Kovach R, George JC, Patlola R, Metzger DC, Mena-Hurtado C, Beasley R, Soukas P, Colon-Hernandez PJ, Stark MA, Walker C; EXCITE ISR Investigators. Randomized controlled study of excimer laser atherectomy for treatment of femoropopliteal in-stent restenosis: initial results from the EXCITE ISR trial (EXCImer Laser Randomized Controlled Study for Treatment of FemoropopliTEal In-Stent Restenosis). JACC Cardiovasc Interv. 2015 Jan;8(1 Pt A):92-101. doi: 10.1016/j.jcin.2014.09.009. Epub 2014 Dec 10. PMID 25499305
- [Background] Shammas NW. JETSTREAM Atherectomy: A Review of Technique, Tips, and Tricks in Treating the Femoropopliteal Lesions. Int J Angiol. 2015 Jun;24(2):81-6. doi: 10.1055/s-0034-1390083. PMID 26060377
- [Derived] Shammas NW, Petruzzi N, Henao S, Armstrong EJ, Shimshak T, Banerjee S, Latif F, Eaves B, Brothers T, Golzar J, Shammas GA, Jones-Miller S, Christensen L, Shammas WJ. JetStream Atherectomy for the Treatment of In-Stent Restenosis of the Femoropopliteal Segment: One-Year Results of the JET-ISR Study. J Endovasc Ther. 2021 Feb;28(1):107-116. doi: 10.1177/1526602820951916. Epub 2020 Sep 4. PMID 32885736

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | JetStream XC With Balloon Angioplasty
Started | 60
Completed | 52 (8 Deaths)
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | JetStream XC With Balloon Angioplasty
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 38
Age, Continuous [Mean (Full Range); unit: years] | 70.2 [49 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 40
Race/Ethnicity, Customized [Number; unit: participants]
  white | 51
  Hispanic | 1
  African American | 8
Region of Enrollment [Number; unit: participants]
  United States | 60
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.4 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Target Lesion Revascularization (TLR)
Description: TLR is defined as retreatment of the index lesion (extended 1 cm proximal and distal to the lesion) at 6 months. For the primary endpoint, intra-procedural bail out stenting of the index lesion is considered meeting a TLR endpoint. (ITT analysis)
Time Frame: 6 months
Population: 5 people died at 6 months. 1 patient had TLR before death and was counted in the TLR analysis. 4 patients were not analyzed at 6 months as they were dead before a TLR occurred (censored). So these 4 patients were excluded from the analysis at 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | JetStream XC With Balloon Angioplasty
Number analyzed (Participants) | 56
Participants | 12

2. Primary Outcome: Major Adverse Events (MAE)
Description: unplanned major amputation, all cause mortality, and Bailout Stenting consider Target Lesion Revascularization (TLR).
Time Frame: 30 days
Population: All patients were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | JetStream XC With Balloon Angioplasty
Number analyzed (Participants) | 60
Participants | 6

3. Secondary Outcome: Device Outcome
Description: Categorized by < 50% residual stenosis following JS atherectomy alone and without additional adjunctive PTA or bail out procedures as determined by the Angiographic Core Laboratory.
Time Frame: Intraprocedural
Population: 15 patients did not have interpretable angiographic films by core lab
Measure: Count of Participants; unit: Participants
Arm/Group | JetStream XC With Balloon Angioplasty
Number analyzed (Participants) | 45
Participants | 25

4. Secondary Outcome: Procedural Success
Description: Defined as ≤30% residual diameter stenosis following JS + PTA without provisional or bailout procedures
Time Frame: Intraprocedural
Population: 11 patients with angiogram not interpretable by core lab
Measure: Count of Participants; unit: Participants
Arm/Group | JetStream XC With Balloon Angioplasty
Number analyzed (Participants) | 49
Participants | 35

5. Secondary Outcome: Target Lesion Revascularization (TLR) With no Bailout Stent Included
Description: TLR is defined as retreatment of the index lesion (extended 1 cm proximal and distal to the lesion) at 6 months. Intra-procedural bail out stenting of the index lesion is NOT considered meeting a TLR endpoint. (ITT analysis)
Time Frame: 6 months
Population: 5 patients died after hospital discharge out of 60 patients
Measure: Count of Participants; unit: Participants
Arm/Group | JetStream XC With Balloon Angioplasty
Number analyzed (Participants) | 55
Participants | 6

6. Secondary Outcome: Target Lesion Revascularization (TLR)
Description: TLR is defined as retreatment of the index lesion (extended 1 cm proximal and distal to the lesion) at 1 year ITT (bail out stent in the Lab is not considered as TLR)
Time Frame: 1 year
Population: 8 patients died at 1 year before TLR occurred and so censored out.
Measure: Count of Participants; unit: Participants
Arm/Group | JetStream XC With Balloon Angioplasty
Number analyzed (Participants) | 52
Participants | 18

7. Secondary Outcome: Clinical Patency
Description: Defined as PSVR ≤ 2.5 at the treated site or < 50% stenosis by angiography as determined by the Angiographic Core Laboratory in the absence of TLR, amputation, and/or surgical bypass (the evaluation of patency is extended to one cm proximal and one cm distal to the target lesion)
Time Frame: 6 months
Population: 20 patients either died or had no duplex US at 6 month to assess patency
Measure: Count of Participants; unit: Participants
Arm/Group | JetStream XC With Balloon Angioplasty
Number analyzed (Participants) | 40
Participants | 31

8. Secondary Outcome: Clinical Patency
Description: as for outcome 7
Time Frame: 1 year
Population: 41 patients either died or did not have a Duplex Ultrasound to assess for patency at 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | JetStream XC With Balloon Angioplasty
Number analyzed (Participants) | 29
Participants | 15

9. Secondary Outcome: Change in Walking Impairment Questionnaire Score
Description: Defined as the change in mean Walking Impairment Questionnaire (WIQ) score at 6 months minus baseline. WIQ score range is 0 to 56. A higher score means a better outcome. WIQ is reported as a change between baseline and 6 months in the score (WIQ score at 6 months minus WIQ score at baseline)
Time Frame: Baseline and 6 months
Population: Data not available on 12 patients that either died or test not performed
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | JetStream XC With Balloon Angioplasty
Number analyzed (Participants) | 48
score on a scale | 21.8 [12.9 to 34.5]

10. Secondary Outcome: Number of Participants With Rutherford Clinical Category Improvement
Description: Defined as the change in clinical status indicated by the number of participants that had one improvement of their Rutherford Becker category by at least 1 category at 6 months. The Rutherford category is done on a scale of 0 (no symptoms) to 6 (gangrene/ulceration). A change downward from one category to another is considered an improvement.
Time Frame: 6 months
Population: 38/49 77.5% participants showed improvment by at least 1 category at 6 months
Measure: Number; unit: participants
Arm/Group | JetStream XC With Balloon Angioplasty
Number analyzed (Participants) | 49
participants | 38

11. Secondary Outcome: Change in Ankle-Brachial Index
Description: Defined as the mean ankle-brachial index (ABI) at 6 months minus mean ABI at baseline in subjects with compressible arteries and baseline ABI < 0.9 (0 to 1.2 is the scale ranging from severe disease to normal respectively; higher is better).
Time Frame: 6 months
Population: The change in ABI at 6 months is a mean of 0.2+/- 0.3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | JetStream XC With Balloon Angioplasty
Number analyzed (Participants) | 38
units on a scale | 0.2 (0.3)

12. Secondary Outcome: Change in Walking Impairment Questionnaire at 1 Year
Description: Defined as the change in mean Walking Impairment Questionnaire (Score 0 to 56. A higher score means a better outcome) from Baseline minus at one Year.
  29.2-48.8 is the confidence interval minimum and maximum values.
Time Frame: 1 Year
Population: 38.7 % improvement from baseline to 1 year.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JetStream XC With Balloon Angioplasty
Number analyzed (Participants) | 43
score on a scale | 38.7 (10.0)

13. Secondary Outcome: Rutherford Clinical Category
Description: Defined as the change in clinical status indicated by the change in Rutherford Becker Class at 1 Year compared to baseline by at least one category that is attributable to the treated limb (in cases of bilateral disease).
  Categories are 0 which is asymptomatic to 6 which is gangrene. (Rutherford Becker Category:0=Asymptomatic, 1 = Mild Claudication, 2=moderated claudication, 3= severe claudication, 4= resting pain, 5= ulcers, 6= ulcers with gangrene.
Time Frame: 1 Year
Population: 17 patients either died or Rutherford Category was not assessed due to no office visit or not evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | JetStream XC With Balloon Angioplasty
Number analyzed (Participants) | 43
Participants | 35

14. Secondary Outcome: Ankle Brachial Index
Description: Defined as the change in mean ankle-brachial index (ABI) at 1 Year minus mean ABI at baseline in subjects with compressible arteries and baseline ABI < 0.9. Units on a Scale: 0 to 1.2 (worse to normal respectively)
Time Frame: 1 Year
Population: 29 patients missing because of death or ABI not obtained at visit or visit did not occur
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | JetStream XC With Balloon Angioplasty
Number analyzed (Participants) | 31
units on a scale | 0.2 [0.2 to 0.3]

15. Secondary Outcome: Clinically Driven Target Lesion Revascularization
Description: Clinically-driven TLR (CD-TLR) at 6 months was defined as any reintervention or bypass graft surgery involving a target lesion with a ≥70% diameter stenosis by angiography or PSVR >3.5 and at least 2 of the following associated events: ≥1-level worsening of the Rutherford category, worsening WIQ score by ≥20 points, or an ABI drop >0.15 between baseline and follow-up.
Time Frame: 6 months
Population: 8/45 experienced CD TLR (by KM)
Measure: Count of Participants; unit: Participants
Arm/Group | JetStream XC With Balloon Angioplasty
Number analyzed (Participants) | 45
Participants | 8

16. Secondary Outcome: Clinically Driven Target Lesion Revascularization
Description: Clinically-driven TLR (CD-TLR) was defined as any reintervention or bypass graft surgery involving a target lesion with a ≥70% diameter stenosis by angiography or PSVR >3.5 and at least 2 of the following associated events: ≥1-level worsening of the Rutherford category, worsening WIQ score by ≥20 points, or an ABI drop >0.15 between baseline and follow-up.
Time Frame: 12 months
Population: 11/32 experienced CD-TLR at 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | JetStream XC With Balloon Angioplasty
Number analyzed (Participants) | 32
Participants | 11

ADVERSE EVENTS:
Time Frame: Major Adverse Events were collected for up to 1 year
Description: Definition are consistent with clinicaltrials.gov definition for AE and SAE
Arm/Group | JetStream XC With Balloon Angioplasty
All-Cause Mortality (participants affected / at risk) | 8/60
Serious Adverse Events (participants affected / at risk) | 21/60
Other Adverse Events (participants affected / at risk) | 15/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JetStream XC With Balloon Angioplasty (N=60)
Target Lesion Revascularization with Bailout Stenting (Vascular disorders) | 21 (21) — Retreatment of the index lesion (extended 1 cm proximal and distal to the lesion). At 1 Year.
Target Lesion Revascularization without Bailout Stenting (Vascular disorders) | 11 (11) — at 1 year
Unplanned Major amputation (Vascular disorders) | 0 (0) — at 1 month
New Stent Fracture or Disruption (Vascular disorders) | 0 (0) — at 1 month
Device Induced Vascular Injury (Vascular disorders) | 0 (0) — at 1 month
Distal Embolization (Vascular disorders) | 8 (8) — at 1 month
Major Bleeding (Blood and lymphatic system disorders) | 1 (1) — at 1 month
Nonfatal myocardial Infarction (Cardiac disorders) | 1 (1) — at 1 month
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JetStream XC With Balloon Angioplasty (N=60)
Angina (Cardiac disorders) | 4 (60) — Chest pain due to ischemic heart disease
worsening claudication in non affected limb (Vascular disorders) | 11 (60) — worsening claudication and interventions on the non affected limb

LIMITATIONS AND CAVEATS:
The built in aspiration system may reduce potential debris, although it does not eliminate this problem completely. Lack of safety data in class III and IV stent fractures and the safety of the device in tortuous vessels (>45 degrees) has not been demonstrated given wire bias in these vessels.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-29): https://cdn.clinicaltrials.gov/large-docs/34/NCT02730234/Prot_SAP_000.pdf